CLINICAL TRIAL: NCT04932798
Title: Genetic Risk-Based Atrial Fibrillation Screening
Brief Title: Genetic Risk-Based Atrial Fibrillation Screening (GeneAF Study)
Acronym: GeneAF
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Julia Cadrin-Tourigny, Cardiologist electrophysiologist, Montreal Heart Institute
Other Study IDs: 2020-2780
Record Dates: First submitted 2021-06-08; First posted 2021-06-21 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Genetic Predisposition; Atrial Fibrillation
MeSH Terms: conditions — Genetic Predisposition to Disease; Atrial Fibrillation | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-Risk group: : Montreal Heart Institute biobank participants with a high specific genome-wide polygenic risk scores for atrial fibrillation G
  Interventions: Diagnostic Test: Resting ECG (if first visit is done on site only); Diagnostic Test: 24-hour ambulatory electrocardiographic monitoring (Holter) (if first visit done on site only); Diagnostic Test: 3-month AF detection monitoring using the Apple Watch
- Low-Risk group: Montreal Heart Institute biobank participants with a low specific genome-wide polygenic risk scores for atrial fibrillation G
  Interventions: Diagnostic Test: Resting ECG (if first visit is done on site only); Diagnostic Test: 24-hour ambulatory electrocardiographic monitoring (Holter) (if first visit done on site only); Diagnostic Test: 3-month AF detection monitoring using the Apple Watch

INTERVENTIONS:
Diagnostic Test: Resting ECG (if first visit is done on site only) — The standard 12-lead electrocardiogram is a representation of the heart's electrical activity recorded from electrodes on the body surface.
  This test requires around 15 minutes of the participant's time.
Diagnostic Test: 24-hour ambulatory electrocardiographic monitoring (Holter) (if first visit done on site only) — The Holter monitor is a type of portable electrocardiogram (ECG) worn continuously for 24 hours.
Diagnostic Test: 3-month AF detection monitoring using the Apple Watch — Patients with irregular heart rates will be notified by the Apple Watch and instructed to confirm the rhythm by using the integrated ECG recording system. This simply requires touching the watch with a finger from the opposite hand and provides a 30 seconds one-lead ECG recording of diagnostic quality. These tracing will be transferred to the study team for analysis using a dedicated email.

SUMMARY:
AF is the most common sustained arrhythmia in adults and its prevalence increases with advancing age.

In this study, we aim to determine whether the published genome-wide polygenic scores for atrial fibrillation (GPSAF) can facilitate AF screening by accurately discriminating between patients with low and high risk for AF.

All included patients are participating in the MHI biobank, an ongoing funded institutional DNA bank and clinical registry approved by the research ethics board where included patients consent for future genetic research.

The study will compare AF detection rate using a 3 months near continuous monitoring in individuals with a high GPSAF with matched individuals from the bottom GPSAF.

DETAILED DESCRIPTION:
In Canada, 50,000 strokes occur every year and can have devastating consequences on patients. Approximately 15% of strokes are attributable to an undiagnosed arrhythmia, atrial fibrillation (AF). Strokes due to AF are more severe and lethal but are preventable with anti-coagulation. Most patients who suffer from AF are asymptomatic and thus don't come spontaneously to medical attention. The diagnosis can be made by electrocardiographical (ECG) recording. As longer recordings spanning on weeks and months are often required, it is not possible to apply this intense screening to the entire population. The GeneAF project thus aims to use genetic information to identify and target patients who benefit the most from a more intensive screening approach. A previously published genetic polygenic risk score (GPS) for AF has been shown to be associated with prevalent AF in the UK biobank population. Participants in the top 5 percentile were three times more likely to have a history of AF (prevalent AF).

The aim of this project is to determine if the use of this previously published GPS score for prevalent AF can be used to screen for silent incident AF in our population.

Primary objective: To assess the association of GPSAF with silent AF and compare AF detection rates in patients with a high GPSAF to matched controls.

Secondary objectives: To determine the proportion of patients with identified AF who will be prescribed anticoagulation during follow-up.

Methods:

The GeneAF study is a cohort study comparing AF detection rate using a 3 months near-continuous monitoring in individuals with a high GPSAF (top 5%; High Risk group) with matched individuals from the bottom 95% GPSAF (Lower Risk group). All included subjects are current participants in the MHI biobank. Only candidates who would be considered for anticoagulation in case AF is detected (actionable AF; CHADS-65 > 1. We estimate that approximately 350 patients per group will be needed.

ELIGIBILITY:
Inclusion Criteria:

* Having a CHADS65 score>1, which requires either:

Age >= 65 and/or A prior Stroke or TIA and/or Hypertension and/or A history of heart failure and/or Diabetes

Exclusion Criteria:

1. Already on oral anticoagulation
2. Any prior history of AF or atrial flutter (AFl)
3. Patients currently having an implantable device (pacemaker, defibrillator or loop recorder) that allows detection of AF/AFl
4. Refusing testing with the "Apple Watch"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included subjects are current participants in the Montreal Heart Institute (MHI) biobank. Only candidates who would be considered for anticoagulation in case atrial firbrillation is detected (actionable AF; CHADS65 > 1) will be considered for inclusion. MHI biobank participants that are eligible for the current study will be contacted to be part of the study.
Sampling Method: Probability Sample
Enrollment: 726 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Detection of atrial fibrillation/atrial flutter (Y/N) | 3 months
  Atrial Fibrillation will be diagnosed according to the standard definition: "at least one 30-second recording with irregular rhythm without p waves". This will be accomplished either through the baseline ECG, Holter or during the 3 months monitoring with the Apple watch.
  The diagnostic of AF with the "Apple watch" requires:
  1. Detection of irregular heart rate (photopletysmography)
  2. Confirmation of the rhythm with a real time single lead 30 seconds ECG with the Apple Watch.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Cadrin-Tourigny, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khera AV, Chaffin M, Aragam KG, Haas ME, Roselli C, Choi SH, Natarajan P, Lander ES, Lubitz SA, Ellinor PT, Kathiresan S. Genome-wide polygenic scores for common diseases identify individuals with risk equivalent to monogenic mutations. Nat Genet. 2018 Sep;50(9):1219-1224. doi: 10.1038/s41588-018-0183-z. Epub 2018 Aug 13. PMID 30104762
- [Background] Wunnemann F, Sin Lo K, Langford-Avelar A, Busseuil D, Dube MP, Tardif JC, Lettre G. Validation of Genome-Wide Polygenic Risk Scores for Coronary Artery Disease in French Canadians. Circ Genom Precis Med. 2019 Jun;12(6):e002481. doi: 10.1161/CIRCGEN.119.002481. Epub 2019 Jun 11. PMID 31184202
- [Background] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151